CLINICAL TRIAL: NCT06062186
Title: Acute Effects of Naturally Occurring Tea and Coffee-based Ingredients on Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AFS-04-2023-003
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Change

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 650 mg of placebo, given as two capsules containing maltodextrin
  Interventions: Dietary Supplement: Placebo
- AmaTea Max Guayusa extract (Experimental): 650 mg of AmaTea Guayusa Extract, given as two capsules
  Interventions: Dietary Supplement: AmaTea Guayusa Extract
- Lion's Mane (Experimental): 1000 mg of Lion's Mane, given as two capsules
  Interventions: Dietary Supplement: Lion's Mane

INTERVENTIONS:
Dietary Supplement: Placebo — 650 mg of placebo, given as two capsules containing maltodextrin
  Arms: Placebo
Dietary Supplement: AmaTea Guayusa Extract — 650 mg of AmaTea Guayusa Extract, given as two capsules
  Arms: AmaTea Max Guayusa extract
Dietary Supplement: Lion's Mane — 1000 mg of Lion's Mane, given as two capsules
  Arms: Lion's Mane

SUMMARY:
This study is a double-blind, randomized, three-arm, single-dose, placebo-controlled crossover trial of forty (40) apparently healthy male and female participants. The objective of this study is to assess the effects of AmaTea Max Organic Guayusa Extract and Lion's Mane on cognitive responses including mental clarity, mood, focus, concentration, productivity, anxiety/stress, happiness, and accuracy.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, three-arm, single-dose, placebo-controlled crossover trial of forty (40) apparently healthy male and female participants. The objective of this study is to assess the effects of AmaTea Max Organic Guayusa Extract and Lion's Mane on cognitive responses including mental clarity, mood, focus, concentration, productivity, anxiety/stress, happiness, and accuracy. Since these dietary supplements are on the market for consumer use, it is important to investigate and confirm their potential benefits, comparisons, and safety through further research.

Subjects will attend 4 study visits. During Visit 1, subjects will be screened for participation (i.e., medical history, routine blood work, background baseline diet). During Visits 2, 3 and 4, at 3 time points (pre-ingestion, 60 and 120 minutes post ingestion), participants will complete subjective baseline testing including questionnaires that assess mental clarity, mood, focus, concentration, productivity, anxiety/stress, and the Happiness Scale in addition to completing a series of objective neuropsychological tests (e.g., Go/no-go test, N-back test, Serial Sevens test) to assess cognitive performance. Safety will be monitored via vital signs (heart rate, blood pressure) and adverse events (AE) throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health and able to participate in cognitive performance testing as determined by assessment, medical history and routine blood chemistries.
* Between the of 18 and 50 years of age (inclusive).
* Body Mass Index of 18.5-39.9 (inclusive).
* Body weight of at least 110 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal supine, resting heart rate (<90 per minute).
* Able to provide an adequate blood draw.
* Habitually consumes ≤ 240 mg caffeine/day (equivalent of 3 cups of coffee). Dietary supplementation consistent over one month and able to maintain supplementation throughout study.
* If dietary supplement initiated within the past month, participant is willing to discontinue supplement use followed by a 2-week washout prior to participation in the study.
* Willing to duplicate their previous 24-hour diet, refrain from caffeine for 12 hours, refrain from exercise for 24 hours prior to each trial, and fast for 8 hours prior each of the treatments.

Exclusion Criteria:

* Current smoker or other nicotine use (i.e. vape, patch, etc.).
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g. electrolyte abnormalities, diabetes, thyroid disease, adrenal disease, hypogonadism, short bowel syndrome, diarrheal illnesses, history of colon resection, gastric ulcer, reflux disease, gastroparesis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition or disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* History of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* History of cognitive disorder.
* History of psychiatric disorder.
* Known sensitivity to any ingredient in the test formulations as listed in the Certificates-of-Analysis.
* Women currently pregnant, trying to become pregnant or breastfeeding a child.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoint or place the subject at increased risk of harm if they were to participate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Concentration | Change from baseline to 60 minutes and 120 minutes.
  Concentration as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent better concentration.
Mental Clarity | Change from baseline to 60 minutes and 120 minutes.
  Mental clarity as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent better mental clarity.
Mood | Change from baseline to 60 minutes and 120 minutes.
  Mood as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent better mood.
Focus | Change from baseline to 60 minutes and 120 minutes.
  Focus as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent better focus.
Productivity | Change from baseline to 60 minutes and 120 minutes.
  Productivity as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent better productivity.
Stress | Change from baseline to 60 minutes and 120 minutes.
  Stress as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent greater stress.
Happiness | Change from baseline to 60 minutes and 120 minutes.
  Happiness as measured by The Subjective Happiness Scale, where values can range from 4 to 28, and higher values represent greater happiness.
Cognitive Control | Change from baseline to 60 minutes and 120 minutes.
  Cognitive control as measured by the Go/No-go Test.
Working Memory | Change from baseline to 60 minutes and 120 minutes.
  Working memory as measured by the N-back Test.
Attention | Change from baseline to 60 minutes and 120 minutes.
  Attention as measured by the Serial Sevens Test.

SECONDARY OUTCOMES:
Systolic blood pressure | Change from baseline to 60 minutes and 120 minutes.
  Systolic blood pressure in mm of mercury.
Diastolic blood pressure | Change from baseline to 60 minutes and 120 minutes.
  Diastolic blood pressure in mm of mercury.
Heart rate | Change from baseline to 60 minutes and 120 minutes.
  Heart rate measured in beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ziegenfuss, PhD, Principal Investigator — The Center for Applied Health Sciences
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided